CLINICAL TRIAL: NCT06672939
Title: Efficacy, Safety, and Pharmacokinetics of Orforglipron Once Daily Oral Versus Placebo in Adolescent Participants Who Have Obesity, or Overweight With Weight-Related Comorbidities: A Randomized, Double-Blind Trial (ADVANCE-ATTAIN-ADOLESCENTS)
Brief Title: A Study of Orforglipron (LY3502970) in Adolescent Participants With Obesity, or Overweight With Related Comorbidities
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18868; J4M-MC-PW01 (Other: Eli Lilly and Company); J4M-MC-PWMP Master Protocol (Other: Eli Lilly and Company); 2024-514081-40-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orforglipron (Experimental): Participants will receive orforglipron orally
  Interventions: Drug: Orforglipron
- Placebo (Placebo Comparator): Participants will receive placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970
  Arms: Orforglipron
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study, performed under Master Protocol J4M-MC-PWMP, is to evaluate the efficacy, safety, and pharmacokinetics of orforglipron once daily oral versus Placebo in adolescent participants with obesity, or overweight with related comorbidities. Participation in the study will last about 18 months.

ELIGIBILITY:
Inclusion Criteria:

J4M-MC-PWMP

* Have a history of at least 1 unsuccessful effort to lose sufficient body weight after participation in a structured lifestyle modification program (diet and exercise counseling for at least 3 months) prior to screening.
* Obesity as defined by BMI equal to or above the 95th percentile for age and sex (on age- and gender-specific growth chart [CDC-NCHS, 2022]); OR
* Overweight as defined by BMI equal to or above the 85th percentile but less than the 95th percentile for age and sex, on age- and sex-specific growth chart (CDC-NCHS, 2022), and at least 1 weight-related comorbidity,

  * hypertension
  * type 2 diabetes (T2D)
  * prediabetes
  * dyslipidemia
  * obstructive sleep apnea
  * metabolic dysfunction-associated steatohepatitis (MASH) or metabolic dysfunction-associated steatotic liver disease (MASLD)

Exclusion Criteria:

J4M-MC-PW01

* Prepubertal (Tanner stage 1)
* Have a self-reported, or by parent or legal guardian where applicable, decrease in body weight greater than 5 kilograms (kg) (11 pounds) within 90 days before screening

J4M-MC-PWMP

* Have undergone or plan to undergo weight reduction procedure during the study, such as, but not limited to:

  * gastric bypass
  * sleeve gastrectomy
  * restrictive bariatric surgery, such as Lap-Band® gastric banding, or
  * any other procedure intended to result in weight reduction.
* Have a diagnosis that is a secondary cause of obesity or have a history of abrupt onset of obesity suggesting a secondary cause, such as hypothalamic, monogenetic, syndromic, or endocrine causes.
* Have type 1 diabetes or history of ketoacidosis, or hyperosmolar state.
* Have HbA1c >9.0% (75 mmol/mol) as measured by central laboratory at screening.
* Have a family or personal history of medullary thyroid carcinoma or Multiple Endocrine Neoplasia Syndrome Type 2.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Mass Index (BMI) | Baseline, Week 72

SECONDARY OUTCOMES:
Change from Baseline in BMI | Baseline, Week 72
Change from Baseline in Body Weight | Baseline, Week 72
Change from Baseline in Waist Circumference | Baseline, Week 72
Change from Baseline in Body Weight Percentile | Baseline, Week 72
  Based on sex- and age-specific growth charts
Change in Impact of Weight on Quality of Life (IWQOL)-Kids Total and Domain Scores | Baseline, Week 72
  The IWQOL-Kids is a validated, 27-item, patient reported outcomes instrument that assesses weight-related quality of life for youth aged 11 to 19 years in 4 domains:
  * physical comfort (6 items)
  * body esteem (9 items)
  * social life (6 items), and
  * family relations (6 items). It has a recall period of "the past 7 days." All items are rated on a 5-point truth scale ("always true" to "never true"). The 4-domain scores and total score range from 0 to 100, with higher scores indicating better quality of life.
Change from Baseline in Systolic Blood Pressure | Baseline, Week 72
Change from Baseline in Diastolic Blood Pressure | Baseline, Week 72
Percent Change from Baseline in Total Cholesterol | Baseline, Week 72
Change from Baseline in Fasting Glucose | Baseline, Week 72
Percent Change from Baseline in Fasting Insulin | Baseline, Week 72
Percent Change from Baseline in Total Body Fat Mass as Determined by Dual-Energy X-Ray Absorptiometry (DXA) | Baseline, Week 72
Pharmacokinetics (PK): Steady State Area Under the Concentration Time Curve (AUC) of Orforglipron | Baseline, Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- United States (15):
  - Carey Chronis MD Pediatric, Infant and Adolescent Medicine, Ventura, California
  - Yale School of Medicine - Yale Diabetes Center (YDC)) Trials, New Haven, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Children's Healthcare of Atlanta - Center for Advanced Pediatrics, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Velocity Clinical Research, Lafayette, Louisiana
  - MedPharmics, LLC, Gulfport, Mississippi
  - Sundance Clinical Research, St Louis, Missouri
  - Lucas Research, Inc., Morehead City, North Carolina
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Health One Hundred Oaks, Nashville, Tennessee
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Houston, Texas
  - La Providence Pediatrics Clinic - Chemidox Clinical Trials, Houston, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - Velocity Clinical Research, Salt Lake City, South Jordan, Utah
- Israel (3):
  - Shamir Medical Center, Beer Jacob
  - Shaare Zedek Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Italy (4):
  - Azienda Ospedaliero Universitaria Meyer, Florence
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento, Verona
- Japan (4):
  - Saitama Medical University Hospital, Iruma-Gun
  - Osaka City General Hospital, Osaka
  - Sagaekiminami Clinic, Saga
  - Shikoku Medical Center for Children and Adults, Zentsujichó
- Poland (4):
  - Krakowskie Centrum Medyczne - FutureMeds, Krakow
  - FutureMeds - Targowek, Warsaw
  - Instytut Diabetologii - Warsaw, Warszewo
  - FutureMeds sp. z o. o., Wroclaw
- United Kingdom (7):
  - Barnsley Hospital NHS Foundation Trust, Barnsley
  - Bristol Royal Hospital for Children, Bristol
  - Addenbrookes Hospital, Cambridge
  - Ninewells Hospital, Dundee
  - Northwick Park Hospital, Harrow
  - Hull Royal Infirmary, Hull
  - Alder Hey Children's Hospital, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Orforglipron (LY3502970) in Adolescent Participants with Obesity, or Overweight with Related Comorbidities — https://trials.lilly.com/en-US/trial/551535